CLINICAL TRIAL: NCT00421174
Title: A Randomized Double-Blind, Placebo-Controlled Trial of Soluble Tumor Necrosis Factor Receptor: Enbrel (Etanercept) for the Treatment of Acute Idiopathic Pneumonia Syndrome Following Allogeneic Cell Transplantation (BMTCTN0403)
Brief Title: Effectiveness of Etanercept for Idiopathic Pneumonia Syndrome Following Stem Cell Transplantation (BMT CTN 0403)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMTCTN0403; BMTCTN0403 (Other: Blood and Marrow Transplant Clinicial Trials Network); U01HL069294-05 (NIH); 465 (Other: BMT CTN)
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2017-08

CONDITIONS: Pneumonia; Idiopathic Pneumonia Syndrome
Keywords: Etanercept; IPS
MeSH Terms: conditions — Pneumonia | interventions — Etanercept; Adrenal Cortex Hormones; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Etanercept (Experimental): Etanercept plus corticosteroids
  Interventions: Drug: Etanercept
- Placebo (Active Comparator): Placebo plus Corticosteroids
  Interventions: Drug: Placebo plus corticosteroid

INTERVENTIONS:
Drug: Etanercept — Etanercept will be given eight doses of study drug over a 4-week period. The initial dose of etanercept will be administered intravenously on Day 0, with subsequent doses administered subcutaneously (SQ). Dosing will be administered twice weekly over 4 consecutive weeks. Additionally, patients in both arms will receive corticosteroids (2 mg/kg/day) Day 0 through Day 7, with subsequent taper as clinically indicated.
  Other Names: Enbrel®
  Arms: Etanercept
Drug: Placebo plus corticosteroid — Patients will receive a total of eight doses of placebo over a 4-week period. The initial dose of placebo will be administered intravenously on Day 0, with subsequent doses administered subcutaneously (SQ). Dosing will be administered twice weekly over 4 consecutive weeks. The placebo will be the inert diluent used for the etanercept formulation.
  Additionally, patients in both arms will receive corticosteroids (2 mg/kg/day) Day 0 through Day 7, with subsequent taper as clinically indicated.
  Other Names: Methylprednisolone
  Arms: Placebo

SUMMARY:
The study is designed as a Phase III, multi-center randomized, double-blind, placebo-controlled trial investigating the use of etanercept for the treatment of acute, non-infectious pulmonary dysfunction (IPS) occurring after allogeneic hematopoietic cell transplantation (HCT).

DETAILED DESCRIPTION:
BACKGROUND:

Over the last two decades, allogeneic hematopoietic cell transplantation (HCT) has emerged as an important treatment for a number of malignant and non-malignant disorders. Unfortunately, several complications, including graft-versus-host disease (GVHD) and pulmonary dysfunction, limit the utility of this aggressive form of therapy. Infectious and non-infectious lung complications occur in 25% to 55% of HCT recipients and account for up to 50% of transplant-related mortality. In about half of affected patients, no infectious organisms are identified in the lungs. Two major types of non-infectious pulmonary injury are recognized: acute idiopathic pneumonia syndrome (IPS) and sub-acute lung injury (obstructive airway disease or bronchiolitis obliterans [BrOb] and restrictive lung disease). The current study will examine the use of etanercept in patients with IPS.

DESIGN NARRATIVE:

Eligible patients will be randomized to receive one of two arms of therapy: (A) etanercept plus corticosteroids, or (B) placebo plus corticosteroids. Patients will receive a total of eight doses of etanercept (or placebo) over a 4-week period. The initial dose of etanercept (or placebo) will be administered intravenously on Day 0, with subsequent doses administered subcutaneously (SQ). Dosing will be administered twice weekly over 4 consecutive weeks. The placebo will be the inert diluent used for the etanercept formulation.

Additionally, patients in both arms will receive corticosteroids (2 mg/kg/day) Day 0 through Day 7, with subsequent taper as clinically indicated. Chest radiographs shall be obtained weekly through Day 28. Plasma cytokine profiles will be obtained on Days 0, 7, and 28.

For patients < 30 days post-transplant: If the patient's clinical condition is such that a broncho-alveolar lavage (BAL) is deemed "not possible to be performed" by the treating physician (or pulmonologist), then the "on study" BAL may be waived. In such circumstances, the patient may register and be randomized to study therapy without the BAL being undertaken.

For patients not on mechanical ventilation: If a BAL is not done, appropriate virology studies on a nasal swab (or nasal washing) are required as a minimum procedure to study entry.

For patients on mechanical ventilation: Microbiologic studies of a deep endotracheal aspirate are allowed in lieu of a formal bronchoscopy procedure. However, no protocol-specified biologic studies (see Section 4.4) will be done on these specimens.

For patients 31-180 days post-transplant: An "on study" bronchoscopy is required in all cases.

If, at any point following initiation of study drug therapy, previously obtained BAL fluid cultures or other BAL fluid analysis become positive for an infectious pathogen, study drug therapy shall be discontinued at that point, and not re-instituted. The patient will discontinue study drug therapy, but will still be followed for outcome.

The primary study endpoint is response at Day 28. Patients who discontinue study drug therapy for any reason will still be followed for primary and secondary study endpoints.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling the following criteria will be eligible for registration in this study:

* Recipient of an allogeneic bone marrow, cord blood, or peripheral blood stem cell transplant. There are no restrictions based upon underlying disease, donor source, degree of human leukocyte antigen (HLA) match, intensity of the pre-transplant conditioning regimen, or the use of a prior donor leukocyte infusion
* Evidence of acute lung injury, based upon the presence of bilateral pulmonary infiltrates (on chest radiograph) and a supplemental oxygen requirement
* No more than 180 days post transplant

Patients fulfilling the following criteria will be eligible for random assignment in this study:

* BAL fluid negative for pathogenic microorganisms as assessed by gram stain and fungal stain
* BAL fluid negative for pathogenic microorganisms, or test result pending, as assessed by the following tests:

  1. Acid fast bacilli stain (AFB)
  2. Bacterial culture (a quantitative culture of at least 10(4) CFU/mL is considered positive)
  3. Viral cultures for respiratory pathogens, including Respiratory syncytial virus (RSV), adenovirus, parainfluenza, influenza A and B, and Cytomegalovirus (CMV)
  4. Fungal and mycobacterial cultures
  5. Pneumocystis carinii pneumonia (PCP) assay, by polymerase chain reaction (PCR), direct fluorescent antibody (DFA) stain, or cytology (per institutional guidelines)

Exclusion Criteria:

* Sepsis syndrome or hypotension in which inotropic support (excluding dopamine of no more than 5 mcg/kg/minute) is required
* Bacteremia within 48 hours prior to study registration
* Documented invasive fungal or systemic viral infection (excluding asymptomatic viruria) within 14 days prior to study registration
* Evidence of CMV infection, based upon an abnormal PCR assay, antigenemia assay, or shell vial culture within 14 days of study registration
* On mechanical ventilation for more than 48 hours at study registration
* Evidence of congestive heart failure by clinical assessment
* Participating in other investigational studies (Phase I, II, or III) for the treatment of acute GVHD within 7 days of study registration (patients enrolled in BMT CTN 0302 are ineligible for study entry)
* Received etanercept within 14 days prior to study registration
* Pregnant or breastfeeding
* On more than 2 mg/kg/day of methylprednisolone equivalent for more than 48 hours, within 7 days prior to study registration
* Known hypersensitivity to etanercept
* History of active tuberculosis (TB) infection
* History of chronic active hepatitis B or hepatitis C infection
* Patients who have undergone a BAL within 72 hours of study registration are ineligible if the BAL fluid is known to be positive for pathogenic microorganisms
* Patients who have relapsed or have developed progressive disease post-transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-08; Primary Completion 2010-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (12):
- United States (12):
  - University of Florida College of Medicine (Shands), Gainesville, Florida
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - DFCI/Partners Cancer Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Yanik GA, Horowitz MM, Weisdorf DJ, Logan BR, Ho VT, Soiffer RJ, Carter SL, Wu J, Wingard JR, Difronzo NL, Ferrara JL, Giralt S, Madtes DK, Drexler R, White ES, Cooke KR. Randomized, double-blind, placebo-controlled trial of soluble tumor necrosis factor receptor: enbrel (etanercept) for the treatment of idiopathic pneumonia syndrome after allogeneic stem cell transplantation: blood and marrow transplant clinical trials network protocol. Biol Blood Marrow Transplant. 2014 Jun;20(6):858-64. doi: 10.1016/j.bbmt.2014.02.026. Epub 2014 Mar 7. PMID 24607553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from September 2007 to August 2011 from 12 different sites.
Period: Overall Study
Arm/Group | Etanercept | Placebo
Started | 18 | 19
Completed | 16 | 18
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Ineligible due to infection | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Median (Full Range); unit: years] | 47.7 [22.9 to 70.1] | 46.4 [21.8 to 68.8] | 46.6 [21.8 to 70.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 8 | 8 | 16
Primary Disease [Number; unit: participants]
  Acute Myelogenous Leukemia (AML) | 1 | 9 | 10
  Myelodysplastic Syndrome (MDS) | 2 | 2 | 4
  Acute Lymphoblastic Leukemia (ALL) | 3 | 4 | 7
  Lymphoma | 3 | 0 | 3
  Other | 7 | 3 | 10
Karnofsky Performance [Number; unit: participants] — Assesses patient self-perceived global quality of life and functioning (excellent = 100, good = 70-90, fair = 50-60, poor < 50), where 100 equals perfect quality of life.
  participants
    70 - 90 | 3 | 1 | 4
    50 - 60 | 5 | 5 | 10
    < 50 | 5 | 10 | 15
    Unknown | 3 | 2 | 5
Conditioning Regimen [Number; unit: participants]
  Myeloablative | 9 | 11 | 20
  Non-myeloablative | 7 | 7 | 14
Recipient Cytomegalovirus Status [Number; unit: participants]
  Positive | 8 | 10 | 18
  Negative | 8 | 7 | 15
  Unknown | 0 | 1 | 1
Total Bilirubin [Median (Full Range); unit: mg/dl] — Serum total bilirubin (mg/dl) at study entry.
  mg/dl | 1.2 [0.2 to 18.9] | 0.9 [0.2 to 10.7] | 1.0 [0.2 to 18.9]
Creatinine [Median (Full Range); unit: mg/dl] — Serum creatinine (mg/dl) at study entry.
  mg/dl | 1.3 [0.6 to 2.5] | 1.4 [0.4 to 2.9] | 1.3 [0.4 to 2.9]
Oxygen Support [Number; unit: participants] — Method of supplemental oxygen support at study entry.
  participants
    Nasal cannula | 10 | 6 | 16
    Face mask | 3 | 5 | 8
    Mechanical ventilation | 2 | 6 | 8
    Unknown | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response will be defined as survival to Day 28 of study, plus discontinuation of all supplemental oxygen support for more than 72 consecutive hours by Day 28.
Time Frame: Day 28
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
percentage of participants | 62.5 [35.4 to 84.8] | 66.7 [41.0 to 86.7]

2. Secondary Outcome: Response to Therapy
Description: Response will be defined as the ability to survive to Day 56 of study, plus the ability to completely discontinue all supplemental oxygen support for > 72 consecutive hours during this time period.
Time Frame: Day 56
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
percentage of participants | 56.3 [29.9 to 80.3] | 50.0 [26.0 to 74.0]

3. Secondary Outcome: Discontinuation of Supplemental Oxygen
Description: The "time required to discontinue supplemental oxygen" will be measured in the number of days from study entry.
Time Frame: Day 56
Measure: Median (Full Range); unit: days
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
days | 9 [1 to 36] | 7 [2 to 30]

4. Secondary Outcome: Corticosteroid Dose
Description: Patients were treated with systemic corticosteroids with methylprednisolone at 2 mg/kg/day on day 0, with taper allowed after day 7.
Time Frame: Day 14 and 28
Measure: Median (Full Range); unit: mg/kg/day
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
mg/kg/day
  Day 14 | 0.94 [0.56 to 1.92] | 1.00 [0.25 to 2.21]
  Day 28 | 0.57 [0.0 to 2.0] | 0.49 [0.03 to 1.04]

5. Secondary Outcome: Overall Survival
Description: Percentage of patients that survived after one year
Time Frame: Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
percentage of participants | 18.8 [6.5 to 46.3] | 16.7 [4.1 to 36.5]

6. Secondary Outcome: Incidence of Infection
Time Frame: Day 56
Measure: Number; unit: Infections
Units Other Than Participants: Total number of infections
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
Number analyzed (Total number of infections) | 20 | 33
Infections
  Bacterial infection | 9 | 21
  Viral infection | 7 | 10
  Fungal infection | 4 | 2

7. Secondary Outcome: Incidence of Toxicity
Time Frame: Day 56
Measure: Number; unit: Toxcities
Units Other Than Participants: Total number of toxicities
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
Number analyzed (Total number of toxicities) | 14 | 25
Toxcities
  Renal | 4 | 3
  Hepatic | 7 | 14
  Cardiac | 1 | 2
  Central nervous system | 2 | 6

8. Secondary Outcome: Incidence of Graft-vs-Host-Disease (GVHD)
Time Frame: Year 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
percentage of participants
  Acute GVHD | 31.2 [11.0 to 58.7] | 44.4 [21.5 to 69.2]
  GVHD | 25.0 [7.3 to 52.4] | 27.8 [9.7 to 53.5]
  Chronic GVHD | 12.5 [1.6 to 38.4] | 0 [0 to 18.5]

9. Secondary Outcome: Incidence of Relapse
Description: Percentage of patients who experience relapse. Deaths without relapse are considered as a competing risk.
Time Frame: Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
Participants | 3 | 2

10. Secondary Outcome: Overall Mortality
Time Frame: Year 2
Measure: Number; unit: participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 16 | 18
participants | 13 | 15

11. Secondary Outcome: Dermatologic Reaction
Time Frame: Day 28
Population: No data collected
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Pro-inflammatory Markers of Pulmonary Disease, in Both BAL Fluid and Plasma
Time Frame: Day 28
Population: No data collected
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1-year post transplant
Description: Serious adverse events are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected adverse events are reported here.
Arm/Group | Etanercept | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=16) | Placebo (N=18)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2010-06-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT00421174/Prot_SAP_ICF_000.pdf